CLINICAL TRIAL: NCT00956267
Title: Letrozole Versus Laparoscopic Ovarian Diathermy for Ovulation Induction in Clomiphene-resistant Women With Polycystic Ovary Syndrome
Brief Title: Letrozole or Laparoscopic Ovarian Diathermy for Women With CC Resistant Polycystic Ovary Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Dr. Hatem Abu Hashim, Associate Prof. of OB/GYN, Mansoura Faculty of Medicine, Mansoura University.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU- 094; FMH-052-K
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; clomiphene resistance; letrozole; Laparoscopic ovarian diathermy
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Letrozole (Experimental): 2.5 mg letrozole oral tablets daily from day 3 of the menses for 5 days up to 6 cycles
  Interventions: Drug: Letrozole
- Laparoscopic ovarian diathermy (LOD) (Active Comparator): Three-puncture technique. Each ovary was cauterized at four points, each for 4 seconds at 40 W for a depth of 4 mm with a mixed current, using an monopolar electrosurgical needle.
  Interventions: Procedure: Laparoscopic ovarian diathermy (LOD)

INTERVENTIONS:
Drug: Letrozole — 2.5 mg letrozole oral tablets daily from day 3 of the menses for 5 days up to 6 cycles
  Arms: Letrozole
Procedure: Laparoscopic ovarian diathermy (LOD) — Three-puncture technique. Each ovary was cauterized at four points, each for 4 seconds at 40 W for a depth of 4 mm with a mixed current, using an monopolar electrosurgical needle.
  Arms: Laparoscopic ovarian diathermy (LOD)

SUMMARY:
The purpose of this study is to compare and determine the efficacy of letrozole administration to that of laparoscopic ovarian diathermy (LOD) in infertile women with Polycystic ovary syndrome(PCOS)not responding to treatment with Clomiphene alone.

DETAILED DESCRIPTION:
In the letrozole group, withdrawal bleeding was achieved using 10 mg of dydrogesterone tablets for 10 days before stimulation, then 2.5 mg of letrozole oral tablets (Femara; Novartis Pharma Services, Switzerland) daily from day 3 of the menses for 5 days up to six cycles. All patients in the control group underwent laparoscopic ovarian diathermy, then followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* CC resistant PCOS

Exclusion Criteria:

* Congenital adrenal hyperplasia
* Cushing syndrome
* Androgen secreting tumors

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Actual)
Dates: Start 2006-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
occurrence of ovulation and midcycle endometrial thickness (mm).

SECONDARY OUTCOMES:
occurrence of pregnancy, miscarriage, multiple pregnancy and live birth rates.

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Abu Hashim, MD. MRCOG, Principal Investigator — Mansoura University Hospital; Abdel Maged Mashaly, MD, Study Director — Mansoura University Hospital; Ahmed Badawy, MD.PhD., Study Chair — Mansoura University Hospital
Locations (1):
- Mansoura University Hospitals,OB/GYN department, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Holzer H, Casper R, Tulandi T. A new era in ovulation induction. Fertil Steril. 2006 Feb;85(2):277-84. doi: 10.1016/j.fertnstert.2005.05.078. PMID 16595197
- [Background] Bayram N, van Wely M, Kaaijk EM, Bossuyt PM, van der Veen F. Using an electrocautery strategy or recombinant follicle stimulating hormone to induce ovulation in polycystic ovary syndrome: randomised controlled trial. BMJ. 2004 Jan 24;328(7433):192. doi: 10.1136/bmj.328.7433.192. PMID 14739186
- [Background] Farquhar C, Lilford RJ, Marjoribanks J, Vandekerckhove P. Laparoscopic 'drilling' by diathermy or laser for ovulation induction in anovulatory polycystic ovary syndrome. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD001122. doi: 10.1002/14651858.CD001122.pub3. PMID 17636653